CLINICAL TRIAL: NCT05261893
Title: Comparative Effects of Elongation Longitudinaux Avec Decoaption Osteo Articulaire and Post Facilitation Stretching Technique in Patients With Knee Osteoarthritis- A Randomized Controlled Trial
Brief Title: Effects of ELDOA Versus Post Facilitation Stretching Technique in Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC-FSD-00252
Record Dates: First submitted 2022-02-20; First posted 2022-03-02 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Knee Osteoarthritis
Keywords: Comparative; Elongation Longitudinaux Avec Decoaption Osteo Articulaire; Post Facilitation Stretching Technique; Knee Osteoarthritis; Randomized Control Trial
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elongation Longitudinaux Avec Decoaption Osteo Articulaire (Experimental): In this we will use myofascial stretching Elongation Longitudinaux Avec Decoaption Osteo Articulaire for knee osteoarthritis. Each patient perform half kneeling posture with homolateral foot and knee in alignment with hip while knee flex to 90° and retrovulsion of the pelvis. Chin tucked in and head towards ceiling. Patient elbow and wrist in extension and arms in external rotation. In this homolateral arm directed anteriorly and pushing arm away from body and contralateral arm directed superiorly and tibia externally rotated.
  This position maintained for 1 minute with 15 secs rest. This group will receive 40 mins of session.
  Interventions: Other: Elongation Longitudinaux Avec Decoaption Osteo Articulaire
- Post Facilitation Stretching (Experimental): This group will receive post facilitation stretching technique. In this all the major muscles of the lower limb (quadriceps, hamstrings ,upper and lower calf muscles) are stretched .And the physiotherapist instruct the patient how to perform stretch . When we target a muscle and perform stretch patient feels sensation of stretch .
  The stretch was hold on to 60 secs and repeated 3 times on each muscle group on each leg.
  Interventions: Other: Post Facilitation Stretching

INTERVENTIONS:
Other: Elongation Longitudinaux Avec Decoaption Osteo Articulaire — It creates tension in the spine and stretch the fascia and is a myofascial stretch technique and manual physical therapy tool
  Arms: Elongation Longitudinaux Avec Decoaption Osteo Articulaire
Other: Post Facilitation Stretching — Post Facilitation Stretching effectively decreases hamstring muscle tightness while also increasing popliteal angle range. Post-facilitation exercise can help to relieve knee pain. It effectively raises ROM or aligns collagen fibers due to the muscle contraction performed immediately before stretching.
  Arms: Post Facilitation Stretching

SUMMARY:
This study aims to assess whether Elongation Longitudinaux Avec Decoaption Osteo Articulaire versus post assistance extending strategy have effects on knee torment. and to check its impact on actual capacity.

DETAILED DESCRIPTION:
A randomized controlled trial will be conducted at Safi Teaching Hospital, Faisal Teaching Hospital and Allied Hospital Fsd after the synopsis has been approved. Patients will be enrolled using a simple random sampling technique. Patients with Knee Osteoarthritis will be chosen based on pre-established inclusion and exclusion requirements. Patients will receive Elongation Longitudinaux Avec Decoaption Osteo Articulaire, and post-facilitation stretching techniques. Two tools will be used to find out the comparison of both groups; Numeric Pain Rating Scale; for knee pain and Lower Extremity Functional Scale; to check the ability of the patient to perform the everyday task and for evaluation of functional impairments for patients with a disorder of lower extremities.

The assessment will need to be done at baseline and follow up will be 15 days after treatment. Each patient will be asked to give their informed consent. Statistical Package of Social Sciences Version 20 will be used for data entry and analysis.

ELIGIBILITY:
Inclusion Criteria:

* It includes both male and female diagnose with knee Osteoarthritis according to history, physical examination and radiological findings and also patient who score more than 3 on Numeric Pain Rating Scale
* Osteoarthritis grade of 3 and lower as determined by using Kallgran and Lawrence Radiographic classification.

Exclusion Criteria:

* If patient is unable to walk or exercise without functional aid and have previous knee surgery.
* Patient with heart condition.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 12th Week
  The Numerical Pain Rating Scale is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0; no pain at all to 10; worst imaginable pain.
Lower Extremity Functional Scale | 12th Week
  The Lower Extremity Functional Scale is a questionnaire containing 20 questions about a person's ability to perform everyday tasks. The LEFS can be used by clinicians as a measure of patients' initial function, ongoing progress and outcome, as well as to set functional goals.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No